CLINICAL TRIAL: NCT00116701
Title: A Study to Evaluate the Efficacy of Converting From Intravenous or Subcutaneous rHuEPO to Intravenous Darbepoetin Alfa (Aranesp®) in Subjects With Chronic Kidney Disease Receiving Haemodialysis
Brief Title: Treatment for Subjects With Chronic Kidney Disease Receiving Haemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040218
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2008-05

CONDITIONS: Kidney Disease
Keywords: Chronic Kidney Disease (CKD); Haemoglobin (Hb); Erthropoetin (EPO); End Stage Renal Disease (ESRD); Recombinant Human Erthropoetic (rHuEPO); Anaemia; Darbepoetin Alfa, Aranesp®; Haemodialysis; Clinical Trial
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp®

SUMMARY:
Treatment period 1:To demonstrate that switching HD subjects with a baseline haemoglobin (Hb) ≥ 10 g/dL and ≤ 13 g/dL from either subcutaneous (SC) or intravenous (IV) rHuEPO to IV darbepoetin alfa results in a mean Hb > 11 g/dL.

Treatment Period 2:To demonstrate that switching subjects with a Hb > 11 g/dL and ≤ 13 g/dL from once weekly IV darbepoetin alfa to once every 2 weeks (Q2W) maintains the mean Hb at > 11 g/dL.

ELIGIBILITY:
Inclusion Criteria: -at least 18 years old - Diagnosis of chronic kidney disease (CKD) and receiving dialysis for at least 3 months prior to screening - Baseline Hb level greater than or equal to 10.0 g/dL and less than or equal to 13.0 g/dL - Adequate iron stores (defined as serum ferritin greater than or equal to 100 µg/L or transferrin saturation [TSAT] greater than or equal to 20%) - Stable IV (epoetin alfa or beta) or SC rHuEPO (epoetin beta) therapy 2 or 3 times per week for at least 8 weeks before screening (stable is defined as less than 25% change in weekly dose and no change in frequency or route) - All subjects must practice adequate contraception (in the judgment of the investigator) throughout this trial. Exclusion Criteria: - Received SC epoetin alfa in the 12 months before screening - Uncontrolled hypertension (diastolic blood pressure greater than 100 mmHg or systolic blood pressure greater than 180 mmHg on 2 separate occasions during screening) - Prior history (within 12 weeks before enrolment) of cardiovascular events including:

* acute myocardial ischemia;
* hospitalization for congestive heart failure;
* myocardial infarction. - Pregnant or breast-feeding women - Treatment with an investigational agent or device within 30 days before screening or scheduled to receive an investigational agent other than those specified by this protocol during the course of this study - Known sensitivity to any of the products to be administered during dosing - Disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-05

PRIMARY OUTCOMES:
Treatment period 1: Mean haemoglobin during the evaluation period (weeks 21-24)
Treatment period 2: Mean haemoglobin during evaluation period 2 (weeks 45-48)

SECONDARY OUTCOMES:
Treatment period 2: Change in Hb between Evaluation Period 1 and Evaluation Period 2
Treatment period 2: The proportion of subjects with a change in Hb between Evaluation Period 1 and Evaluation Period 2 within the inclusive range -1.0 to +1.5 g/dL
Treatment period 2: The proportion of subjects with a mean Hb > 11.0 g/dL during Evaluation Period 2
Treatment period 2: Dose and frequency of darbepoetin alfa administration over the treatment period
Treatment period 1:The proportion of subjects with a mean Hb > 11.0 g/dL during the evaluation period
Treatment period 1: Change in Hb between screening/baseline and the evaluation period
Treatment period 1: Dose and frequency of darbepoetin alfa administration over the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20040218.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/